CLINICAL TRIAL: NCT05156138
Title: The Possible Association Between Pseudoexfoliation Syndrome And Corneal Endothelial Cell Changes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Ashraf Alhussaini, Principal Investigator, Assiut University
Other Study IDs: AssiutUAA
Record Dates: First submitted 2021-11-25; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Pseudoexfoliation Syndrome
Keywords: Pseudoexfoliation syndrome; Corneal endothelial count
MeSH Terms: conditions — Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: patients with pseudoexfoliation fulfilling the inclusion criteria
  Interventions: Other: no interventions as it is a case control observational study
- control group: patients without pseudoexfoliation fulfilling the inclusion criteria
  Interventions: Other: no interventions as it is a case control observational study

INTERVENTIONS:
Other: no interventions as it is a case control observational study — no interventions as it is a case control observational study

SUMMARY:
The study aims to compare the endothelial cell count in patients with pseudoexfoliation syndrome to the the endothelial cell count in normal patients above the age of 50.

DETAILED DESCRIPTION:
Pseudoexfoliation syndrome is a systemic, age related condition, characterized by the deposition of a basement membrane like material within the anterior segment of the eye, most notably on the anterior lens capsule, the iris, the anterior chamber angle, and the anterior vitreous. Both genetic and environmental factors may play a role in its pathogenesis . This condition may present unilaterally or bilaterally and is known to be a major risk factor for secondary open angle glaucoma. Pseudoexfoliation glaucoma is seen in up to 50% of eyes with pseudoexfoliation. In contrast to primary open angel glaucoma, this disease runs a more aggressive clinical course with high intraocular pressure at onset, fast rate of progression, poor the response to medical therapy is, as well as increased need for surgical intervention.

The prevalence of pseudoexfoliation syndrome demonstrates considerable geographic, ethnic and racial variation, ranging from low rates (< 6% in patients older than 70 years) to higher rates (more than 15%) in other regions. In Egypt, the reported incidence of pseudo-exfoliation syndrome in the population older than 40 years of age is 4.14%.

Several studies have shown the influence of pseudoexfoliation syndrome on the corneal endothelium cell density (ECD). Multiple studies showed decreased ECDs of patients with pseudoexfoliation syndrome compared to control patients. However, since the pseudoexfoliation syndrome varies greatly between different populations, in terms of prevalence and progression, it is valuable to study the potential corneal endothelial cell changes in an Egyptian population.

Factors that can change corneal density include Age, race, history of intraocular surgery, use of contact lenses and endothelial dystrophies. That's why in this study, history of intraocular surgery, corneal endothelial dystrophies and contact lens use are among exclusion criteria and includes patients 50 years in age or older.A low endothelial cell count may be a risk in cataract surgery if needed.

ELIGIBILITY:
Inclusion Criteria:

- Pesudoexfoliation Egyptian patients and controls groups must be at least 50 years old and matched from age.

Controls will be selected from the same outpatient clinic.

Exclusion Criteria:

* Patients with history of previous intraocular surgeries, wearing contact lens and endothelial dystrophies.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients above the age of 50 at the outpatient clinic
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-24 (Estimated); Primary Completion 2022-07-24 (Estimated); Study Completion 2022-09-24 (Estimated)

PRIMARY OUTCOMES:
to determine the possible association between pseudoexfoliation syndrome and corneal endothelial cell changes by measuring: | one year
  1. Endothelial cell density by specular microscopy to be categorized qualitatively into one of two groups (normal/abnormal cell count):
     A. A group with normal cell count (2100-3200 cells/mm2) B. A group with low or abnormal cell count (less than the previous range).
  2. Pseudoexfoliation presence: to qualitatively categorize patients into one of two groups (pseudoexfoliation/ No pseudoexfoliation)

SECONDARY OUTCOMES:
Endothelial cell morphology: to qualitatively categorize the patient subjectively into normal and abnormal shape using specular microscopy. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university, Asyut, Egypt